CLINICAL TRIAL: NCT00061061
Title: The Effects of ERT on Appetitive Behavior and Withdrawal in Short-term Smoking Cessation Compared to Smoking ad Lib in Postmenopausal Female Smokers.
Brief Title: Tobacco Cessation in Postmenopausal Women (Part I) - 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08075-1; R01DA008075-01 (NIH)
Record Dates: First submitted 2003-05-21; First posted 2003-05-22 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Tobacco Use Disorder
Keywords: Tobacco Cessation; Postmenopausal Women
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to evaluate the effects of ERT on appetitive behavior and withdrawal in short-term smoking cessation compared to smoking ad lib in postmenopausal female smokers.

DETAILED DESCRIPTION:
Female subjects were screened and randomized. Following two weeks of medication monitoring, all participants continued smoking as usual for one week, at which time baseline measurements were taken. For the remaining two weeks (the experimental period), participants were randomized to a continued smoking or smoking abstinence condition. The abstinent group was provided with cessation counseling and monitored for abstinence. For all participants, data were collected during five clinic visits on all dependent measures: MNWS, QSU, Beck Depression Inventory (BDI), Profile of Mood States, Motor Speed Tasks and Reaction Time Tests. Question of interest was whether hormone replacement therapy would improve these dependent measures as manifested during short-term smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

Female smokers ages 40-79, smoking at least 15 cigarettes per day for at least one year, have natural menopause, have a transvaginal ultrasound to confirm loss of follicular activitiy, have a normal baseline mammogram, a normal chemistry at baseline, willing to take hormone replacement therapy for the duration of the study, normal thyroid function, and have a normal TSH.

Exclusion Criteria:

Women who have had formal dieting with or without pharmacological methods within the last three months; a weight change greater than or equal to 10 pounds within the last three months, BMI greater than or equal to 40, severe menopausal symptoms, active medical problems, alcohol or drug abuse, other forms of nicotine use.

Ages: 40 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0
Dates: Start 1997-03; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Smoking Cessation Outcomes | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Allen, Ph.D., M.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States